CLINICAL TRIAL: NCT06566846
Title: Lumbosacral Transitional Vertebra(LSTV ) Prevalence in Egypt Population and Its Association With Lumbar Degeneration :Retrospective Evaluation of Consecutive Abdominal CT Scans
Brief Title: Lumbosacral Transitional Vertebra Prevalence Among Egypt Population and Its Association With Lumbar Degeneration
Acronym: LSTV
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samaa Mostafa El-kossi, academic lecturer, Assiut University
Other Study IDs: AssuitU12345
Record Dates: First submitted 2024-08-07; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Lumbosacral Anomalies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LSTV group and control group
- 1 and 2: 1. for cases with LSTV
  2. for normal studies

SUMMARY:
retrospective cross sectional study Study Setting: Cases will be recruited from the recorded data system at the department of diagnostic radiology, Assiut University.

DETAILED DESCRIPTION:
* Study subjects:

  1. Inclusion criteria:

     * All patients underwent MSCT KUB from 2022 till 2023
     * Age between 20-50 years old
  2. Exclusion criteria:

     * All cases below 20 and above 50 .
     * previous history of lumbar spine surgery;
     * non-degenerative pathologies in the lumbar spine which could interrupt the evaluation of lumbar spine degeneration, including spinal tumors, infections, and traumatic fractures;
     * images with poor quality
  3. Sample Size Calculation:

     The study will include all patients underwent KUB CT in Assuit university hospital.

     Objective of this research study will be accomplished through the following consecutive steps:
* Patient Enrolment and sample collection:

Sample are patients underwent MSCT KUB at our hospital , ASSUIT university at one year. Lumbosacral spine will be assessed for LSTV ,the patient images will be divided into two groups ,one which has LSTV as cases and other group with normal spine as control. both groups will be assessed for associated disc degeneration ,facet arthropathy sacroiliac joint degeneration ,paravertebral muscle volume and will be compared with control.

ELIGIBILITY:
Inclusion Criteria:

* • All MSCT KUB studies from 2022 till 2023

  * age between 20-50

Exclusion Criteria:

* All cases below 20 and above 50 .
* previous history of lumbar spine surgery;
* non-degenerative pathologies in the lumbar spine which could interrupt the evaluation of lumbar spine degeneration, including spinal tumors, infections, and traumatic fractures;
* images with poor quality

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include all patients underwent KUB CT in Assuit university hospital at one year.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
prevalence | one year
  prevalence of LSTV among egyptians

SECONDARY OUTCOMES:
correlation of LSTV with lumbar disc degeneration | one year
  association between LSTV and disc height ,segmental disc wedge angle and degree of disc prolapse(mild ,moderate ,severe)
correlation of LSTV with facet joint arthropathy | one year
  fact joint arthropathy will be assessed as unilateral ,bilateral and its degree(mild ,moderate ,severe)
correlation of LSTV with sacroiliac degeneration | one year
  sacroiliac joint will be assessed as unilateral ,bilateral and degree (mild ,moderate ,severe)
correlation of LSTV with paravertebral muscle volume | one year
  bilateral psoas muscle volume in cubic centimeter